CLINICAL TRIAL: NCT05958407
Title: A Phase 3b, Interventional, Adaptive, Clinical Trial to Evaluate the Efficacy and Safety of Tralokinumab 300 mg Every Second Week Monotherapy Compared With Placebo in Subjects With Moderate-to-severe Atopic Hand Eczema Who Are Candidates for Systemic Therapy
Brief Title: A 32-week Trial to Evaluate the Efficacy and Safety of Tralokinumab in Subjects With Moderate-to-severe Atopic Hand Eczema Who Are Candidates for Systemic Therapy
Acronym: ADHAND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0162-2328; U1111-1285-7014 (Other: World Health Organization (WHO)); 2022-502653-34-00 (EU CTIS Number)
Record Dates: First submitted 2023-07-13; First posted 2023-07-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis; Atopic Hand Eczema
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tralokinumab (Experimental): Tralokinumab is administered for 32 weeks (16 weeks double-blinded period + 16 weeks open-label period)
  Interventions: Drug: Tralokinumab
- Placebo + tralokinumab (Placebo Comparator): Placebo is administered for 16 weeks (double-blinded period) prior to roll-over to a 16 weeks open-label period where tralokinumab is administered
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tralokinumab — After a loading dose of 600 mg under the skin (s.c.) at baseline, trial participants are administered a dose of 300 mg every two weeks for 32 weeks
  Arms: Tralokinumab
Drug: Placebo — After a loading dose under the skin (s.c.) at baseline, trial participants are administered a placebo dose every two weeks for 16 weeks
  Arms: Placebo + tralokinumab

SUMMARY:
The purpose of this study is to test if treatment with tralokinumab is safe and effectful to treat moderate-to-severe atopic hand eczema. This will be judged by a range of assessments that rate the severity and extent of atopic hand eczema and its symptoms, as well as general health status and quality of life.

The trial will last for up to 40 weeks. There will be up to 15 visits, 3 of which will be conducted by phone. The first part of the trial is called a screening period and will last up to 4 weeks. For the first 16 weeks after screening, trial participants will receive either tralokinumab or dummy injections every two weeks. After the first 16 weeks, all trial participants will receive tralokinumab injections every two weeks for 16 weeks. The last part of the trial is a period of 4 weeks after the end of treatment period, where trial participants are off the drug for safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above at screening
* Diagnosis of atopic dermatitis (AD) as by the Hanifin and Rajka (1980) criteria for AD
* History of AD for ≥1 year
* Presence of atopic hand eczema (AHE) that has persisted for more than 3 months or returned twice or more within the last 12 months, with avoidance of any known and relevant irritants and allergens
* AD involvement of at least one body location other than the hands and wrists at screening
* An Investigator's Global Assessment AHE score of 3 or 4 (moderate to severe) at screening and baseline
* A HESD itch score (weekly average) of ≥4 at baseline
* Subjects who have a documented recent history (within 12 months before the screening visit) of inadequate response to treatment of AHE with topical prescription medications or for whom topical treatments are otherwise medically inadvisable (e.g., due to important side effects or safety risks)

Exclusion Criteria:

* Subjects must not enter the trial if they have active subtypes of hand eczema other than AHE that are considered to be the predominant cause of the current hand eczema including:

  * Active irritant contact dermatitis
  * Active allergic contact dermatitis
  * Active protein contact dermatitis/contact urticaria
  * Active hyperkeratotic hand eczema
  * Active vesicular hand eczema (pompholyx)
* Active dermatologic conditions that may confound the diagnosis of AD or AHE, or that would interfere with the assessment of treatment
* Use of tanning beds or phototherapy (e.g., UVB, UVA1, PUVA), or Grenz ray therapy on the hands or wrists within 28 days prior to baseline or use of bleach baths on the hands or wrists within 7 days prior to baseline
* Treatment with systemic immunosuppressive/immunomodulating drugs and/or systemic corticosteroids within 28 days prior to baseline
* Treatment with topical corticosteroids, topical calcineurin inhibitors, topical phosphodiesterase 4 inhibitors, or topical Janus kinase inhibitors within 7 days prior to baseline
* Receipt of any marketed biological therapy (i.e. immunoglobulin, anti immunoglobulin E) including dupilumab or investigational biologic agents 3 to 6 months prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
IGA-AHE score of 0 (clear) or 1 (almost clear) | At Week 16
  IGA-AHE: The Investigator's Global Assessment for atopic hand eczema (IGA-AHE) is an instrument to rate the severity of the subject's AHE and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).

SECONDARY OUTCOMES:
Having a decrease in HECSI of at least 75% (HECSI-75) | From baseline (Day 1) to Week 16
  HECSI: The Hand Eczema Severity Index (HECSI) is an instrument used in clinical trials to rate the severity of 6 clinical signs using a 4-point severity scale ranging from 0 (none/absent) to 3 (severe) and the extent of the lesions on each of the 5 hand areas by assessing the percentage of the areas these lesions occupy and converting it to a score based on a 5-point scale.
Having a decrease in HECSI of at least 50% (HECSI-50) | From baseline to Week 16
Having a decrease in HECSI of at least 90% (HECSI-90) | From baseline to Week 16
Percentage change in HECSI score | From baseline to Week 16
Having a ≥2-point reduction in IGA-AHE score | From baseline to Week 16
Reduction in HESD itch score (weekly average) of ≥4 points | From baseline to Week 16
  HESD: The Hand Eczema Symptom Diary (HESD) is a 6-item patient-reported outcome where the subject assesses the worst severity of 6 individual signs and symptoms of hand eczema over the past 24 hours using an 11-point numeric rating scale with anchors of 0 ='no (symptom)' and 10 ='severe (symptom)'. Only the items on itch and pain will be completed.
Reduction in HESD pain score (weekly average) of ≥4 points | From baseline to Week 16
  Among subjects with a baseline HESD pain score (weekly average) ≥4 points.
Percentage change in HEIS score | From baseline to Week 16
  HEIS: The Hand Eczema Impact Scale (HEIS) includes 9 items addressing the subject's perception of the impact of hand eczema on their daily activities over the past 7 days. Each item is scored on a 5-point scale (0='not at all', 1='a little', 2='moderately', 3='a lot', 4='extremely').
Percentage change in DLQI score | From baseline to Week 16
  DLQI: The Dermatology Life Quality Index (DLQI) consists of 10 items addressing the subject's perception of the impact of their skin disease on different aspects of their quality of life over the last week. Each item is scored on a 4-point Likert scale (0 = 'not at all ⁄not relevant'; 1 = 'a little'; 2 = 'a lot'; 3 = 'very much').
Percentage change in HESD itch score (weekly average) | From baseline to Week 16
Percentage change in HESD pain score (weekly average) | From baseline to Week 16
Change in WPAI+CIQ:AHE domain scores | From baseline to Week 16
  WPAI+CIQ:AHE: The impact of AHE on the subject's ability to work/school and perform regular activities will be assessed by WPAI+CIQ:AHE, which is an instrument to measure impairments in both paid work and unpaid work/school attendance. The WPAI+CIQ:AHE consists of 10 items, and scores can be calculated for 7 domains, each reflecting the percentage impairment due to AHE during the past 7 days, with higher numbers indicating greater impairment and less productivity/school attendance.
Number of treatment-emergent adverse events | From baseline to Week 16
IGA-AHE score of 0 (clear) or 1 (almost clear) | At Week 32
Having a decrease in HECSI of at least 75% (HECSI-75) | From baseline to Week 32
Reduction in HESD itch score (weekly average) of ≥4 points | From baseline to Week 32
Reduction in HESD pain score (weekly average) of ≥4 points | From baseline to Week 32
  Among subjects with a baseline HESD pain score (weekly average) ≥4 points
Percentage change in HEIS score | From baseline to Week 32
Percentage change in DLQI score | From baseline to Week 32
Change in WPAI+CIQ:AHE domain scores | From baseline to Week 32
Number of treatment-emergent adverse events during the open-label treatment period | Week 16 to Week 32

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (61):
- United States (22):
  - LEO Pharma Investigational Site, Birmingham, Alabama
  - LEO Pharma Investigational Site, Fort Smith, Arkansas
  - LEO Pharma Investigational Site, Fountain Valley, California
  - LEO Pharma Investigational Site, Los Angeles, California
  - LEO Pharma Investigational Site, Sacramento, California
  - LEO Pharma Investigational Site, Farmington, Connecticut
  - LEO Pharma Investigational Site, Hialeah, Florida
  - LEO Pharma Investigational Site, Plainfield, Indiana
  - LEO Pharma Investigational Site, Louisville, Kentucky
  - LEO Pharma Investigational Site, New Orleans, Louisiana
  - LEO Pharma Investigational Site, Bangor, Maine
  - LEO Pharma Investigational Site, Caledonia, Michigan
  - LEO Pharma Investigational Site, Detroit, Michigan
  - LEO Pharma Investigational Site, Portsmouth, New Hampshire
  - LEO Pharma Investigational Site, Cortland, New York
  - LEO Pharma Investigational Site, New York, New York
  - LEO Pharma Investigational Site, Portland, Oregon
  - LEO Pharma Investigational Site, Nashville, Tennessee
  - LEO Pharma Investigational Site, Dallas, Texas
  - LEO Pharma Investigational Site, Frisco, Texas
  - LEO Pharma Investigational Site, San Antonio, Texas
  - LEO Pharma Investigational Site, Webster, Texas
- Belgium (3):
  - LEO Pharma Investigational Site, Brussels
  - LEO Pharma Investigational Site, Edegem
  - LEO Pharma Investigational site, Ghent
- Canada (11):
  - LEO Pharma Investigational Site, Calgary, Alberta
  - LEO Pharma Investigational Site, Edmonton, Alberta
  - LEO Pharma Investigational Site, Red Deer, Alberta
  - LEO Pharma Investigational Site, Surrey, British Columbia
  - LEO Pharma Investigational Site, Fredericton, New Brunswick
  - LEO Pharma Investigational Site, Hamilton, Ontario
  - LEO Pharma Investigational Site, Richmond Hill, Ontario
  - LEO Pharma Investigational Site, Toronto, Ontario
  - LEO Pharma Investigational Site, Windsor, Ontario
  - LEO Pharma Investigational Site, Saint-Jérôme, Quebec
  - LEO Pharma Investigational Site, Québec
- France (3):
  - LEO Pharma Investigational Site, Nantes
  - LEO Pharma Investigational Site, Pierre-Bénite
  - LEO Pharma Investigational Site, Rouen
- Germany (6):
  - LEO Investigational Site, Bretzenheim
  - LEO Pharma Investigational Site, Frankfurt am Main
  - LEO Pharma Investigational Site, Haßfurt
  - LEO Pharma Investigational Site, Osnabrück
  - LEO Pharma Investigational Site, Tübingen
  - LEO Pharma Investigational Site, Wuppertal
- Netherlands (2):
  - LEO Pharma Investigational Site, Amsterdam
  - LEO Pharma Investigational Site, Groningen
- Poland (2):
  - LEO Pharma Investigational Site, Gdansk
  - LEO Pharma Investigational Site, Krakow
- South Korea (5):
  - LEO Pharma Investigational Site, Wŏnju, Gangwon-do
  - LEO Pharma Investigational Site, Ansan-si, Gyeonggi-do
  - LEO Pharma Investigational Site, Yangsan, Gyeongsangnam-do
  - LEO Pharma Investigational Site, Daegu
  - LEO Pharma Investigational Site, Seoul
- Spain (4):
  - LEO Pharma Investigational Site, Badalona, Barcelona
  - LEO Pharma Investigational site, Alicante
  - LEO Pharma Investigational site, Barcelona
  - LEO Pharma Investigational site, Granada
- United Kingdom (3):
  - LEO Pharma Investigational Site, Salford, Greater Manchester
  - LEO Pharma Investigational Site, Middlesbrough, North Yorkshire
  - LEO Pharma Investigational Site, London

IPD SHARING:
Plan to Share IPD: No